CLINICAL TRIAL: NCT05823818
Title: EUropean Real World Outcomes With Pulsed Field AblatiOn in Patients With Symptomatic AtRIAl Fibrillation
Brief Title: EUropean Real World Outcomes With Pulsed Field AblatiOn
Acronym: EU-PORIA
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Sponsor
Other Study IDs: 20230001
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Catheter Ablation — Catheter Ablation of Atrial Fibrillation

SUMMARY:
Background: Real world clinical evidence using pulsed field ablation (PFA) for atrial fibrillation (AF) ablation is still scarce. In particular, data on longer term outcome from multi-center experience is missing.

Aim: To describe real-world adaption, work-flow data as well as procedural and follow-up outcomes after PFA guided AF ablation in early European users.

Methods: A multi-center registry, European real-world outcomes with Pulsed Field Ablation in Patients with Symptomatic AF - EU-PORIA - was designed.

All-comer data of patients with symptomatic atrial fibrillation (AF) who underwent catheter ablation using PFA will be collected from 7 European high-volume centers who were involved in the early market release of the FARAPULSE technology. Data includes patient demographics, procedural metrics on safety and efficacy as well as follow-up outcome data. Learning curve characteristics and comparison on different workflows will be assessed.

DETAILED DESCRIPTION:
Design A retrospective multi center registry will be conducted assessing European Real World Outcomes with Pulsed Field Ablation in Patients with Symptomatic Atrial Fibrillation (EU-PORIA registry). In total, seven high volume PFA centers from Europe will collect data on center characteristics, demographic patient information, procedural metrics, safety and efficacy parameters as well as 12 months clinical outcome with regards to freedom from atrial tachyarrhythmia and major adverse cardiovascular events (MACE).

Inclusion criteria All patients who underwent an AF catheter ablation procedure using the FARAPULSE PFA system until 31.05.2022 will be included into the analysis.

Endpoints The analysis will focus on variable endpoints.

1. Assessment of 6 months and 12 months clinical success rate defined as freedom from use of any Type I or Type III antiarrhythmic medication for the treatment of AF, AFL, or AT after the blanking period.
2. Description of the incidence of major adverse cardiovascular events (MACE) during or after the ablation.
3. Evolution of procedural metrics (procedure time, fluoroscopy time, safety) during the adoption of the technology across different centers and operators.
4. Comparison of different workflows for the PFA ablation procedure and the effects on outcomes.
5. Analysis of repeat ablation procedures after an index PFA ablation with focus on lesion durability and type of arrhythmia recurrence.

Number of Patients It is expected that up to 1500 patients from 7 European centers will enter the registry.

Timeline This is a retrospective study. Data of above defined patients will be collected until January 15th. After database cleaning and plausibility checks statistical analysis will be carried out. To increase the number of patients with 12 M follow-up, another data-update will be performed end of May 2023.

Statistical analysis Descriptive and comparative analyses will be performed using appropriate statistical tests. Kaplan Meier arrhythmia free survival curves using logistic regression analysis will be computed.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent an AF catheter ablation procedure using the FARAPULSE PFA system until 31.05.2022

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic Atrial Fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1233 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Arrhythmia Free Survival | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardioangiologisches Centrum Bethanien, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Futing A, Neven K, Bordignon S, Reichlin T, Blaauw Y, Hansen J, Adelino R, Ouss A, Roten L, Mulder BA, Ruwald MH, Mene R, van der Voort P, Reinsch N, Kueffer T, Boveda S, Albrecht EM, Raybuck JD, Sutton B, Chun KRJ, Schmidt B. Pulsed Field Ablation as First-Line Therapy for Atrial Fibrillation: A Substudy of the EU-PORIA Registry. Circ Arrhythm Electrophysiol. 2024 Dec;17(12):e013088. doi: 10.1161/CIRCEP.124.013088. Epub 2024 Nov 27. PMID 39601122